CLINICAL TRIAL: NCT00755911
Title: Treatment of Alveolar Bone Defects Using Aastrom Biosciences Autologous Tissue Repair Cell Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Vericel Corporation (Industry)
Responsible Party: Principal Investigator, Darnell Kaigler, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-02
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Results first posted 2014-04-15 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-05

CONDITIONS: Alveolar Bone Loss
Keywords: dental; tooth; implant; extraction; Oral; Surgical; Procedures
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Gelatin Sponge, Absorbable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tissue Repair Cells (TRC) (Experimental): Subjects will receive Tissue Repair Cell (TRC) therapy plus Gelfoam carrier
  Interventions: Biological: Tissue Repair Cells (TRC); Device: Control
- Control (Sham Comparator): Subjects will receive the control treatment, consisting of Gelfoam carrier without Tissue Repair Cell (TRC) therapy.
  Interventions: Device: Control

INTERVENTIONS:
Biological: Tissue Repair Cells (TRC) — 30-50 ml of bone marrow is aspirated from subject and processed into TRC autologous bone marrow tissue graft. 10ml of TRC will be absorbed onto gelfoam carrier and placed in extraction socket.
  Other Names: Tissue Repair Cells, Bone Repair Cells, ixmyelocel-t
  Arms: Tissue Repair Cells (TRC)
Device: Control — Control subjects only receive standard gelfoam carrier. It promotes healing after tooth extraction
  Other Names: Gelfoam

SUMMARY:
The purpose of this research is to determine if a subject's own bone marrow tissue can help regenerate bone in the area of his/her jaw where a tooth has been removed using Tissue Repair Cell (TRC) Therapy.

DETAILED DESCRIPTION:
A sample of the subject's bone marrow tissue will be collected and sent to a laboratory where it will be processed to form cells. The new cells are transplanted into the tooth socket after the tooth has been removed. The researchers are testing to see if these cells (TRC) will help form bone. The research will also determine if the implant the subject receives will be more stable in the area with new bone growth.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 20 to 70 years
* Gender: Male and female
* Patients must be able and willing to follow study procedures and instructions
* Patients must have read, understood and signed an informed consent form
* Patients must require tooth extraction as a result of caries, periodontal disease, or tooth fracture

Exclusion Criteria:

* Allergies or hypersensitivities to study related medications: amoxicillin, dexamethasone, chlorhexidine, ibuprofen, ranitidine
* Hematologic disorders/ blood dyscrasias
* Active infectious disease
* Liver or kidney dysfunction/failure- Patients will have blood drawn for serum laboratory tests, including creatinine, blood urea nitrogen (BUN), aspartate aminotransferase (AST), alanine aminotransferase test (ALT), and bilirubin. All of these must be within normal limits for a patient to be included in the study. Current University of Michigan Health System normal lab values are as follows: Creatinine (male 0.7-1.3 mg/dl; female 0.5-1.0 mg/dl); BUN (8-20 mg/dl); AST (8-30 IU/L); ALT (7-35 IU/L); Bilirubin (0.2-1.2 mg/dl).
* Endocrine disorders/dysfunctions (i.e Type I and II diabetes)
* Cancer - The explicit definition of cancer used to exclude patients is consistent with that described by the National Cancer Institute (NCI), National Institutes of Health. According to NCI, cancer is any disease in which abnormal cells divide without control and invade nearby tissues (invasive disease). These include carcinomas, sarcomas, leukemias, and lymphomas. Any patient with a history of these invasive diseases will be excluded from the study.
* Patients who currently use bisphosphonates or have a history of bisphosphonate use will be excluded from the trial.
* HIV+
* Metabolic Bone Diseases-Patients with metabolic bone diseases such as Paget's disease, hypercalcemia, moderate to severe vitamin D3 abnormalities or any other metabolic bone disease including osteoporosis and osteoporotic fractures will be excluded. The following scale will be used to determine osteoporosis in patients who have had a bone mass density (BMD) determination: Normal = T score at or above -1.0 SD; Osteopenia = T score between -1.0 and -2.5 SD; Osteoporosis = T score at or below -2.5 standard deviation (SD). Although a dexa scan will not be required, all post-menopausal women receiving osteoporosis/osteopenia related therapy will receive a dexa scan as part of their standard medical care.
* Additionally, individuals who have a medical history significant for diabetes will not be included in the study.
* Laboratory values that will define normal renal and hepatic function, as well as criteria for exclusion of metabolic bone disease are consistent with those established by the University of Michigan Health System (UMHS). Normal clinical values will be used to help assure the health of all subjects in this trial.
* Individuals who have a BMI outside normal limits or a BMI that deems them overweight (BMI >25) will be excluded due to potential difficulties in locating appropriate surgical entry of the iliac crest during bone marrow aspiration procedure.
* The following additional exclusion criteria for regenerative sites are in alignment with those described and adapted for using bone morphogenetic protein (BMPs) to regenerate buccal wall defects (Fiorellini, Howell et al. 2005):
* Patients < 20 and > 60 years of age
* Pregnant women- Female patients who are of childbearing potential are excluded except those who are using hormonal or barrier methods of birth control (oral or parenteral contraceptives, transdermal patch, diaphragm plus spermicide, or condoms). Pregnancy status will be determined with a urine test and patients who are pregnant, as determined by a positive test, will be excluded from the study
* Patients with acute sinusitis
* Patients with congenital or metabolic bone disorders
* Current smokers (have smoked within 6 mos. of study onset)
* Presence of < 4 mm of bone from apex of tooth to the alveolar crest
* < 2 mm bone from apex to floor of maxillary sinus

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-06; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darnell Kaigler, DDS, MS, PhD, Principal Investigator — University of Michigan Department of Periodontics and Oral Medicine; William V Giannobile, DDS, DMedSc, Study Chair — University of Michigan Center for Oral Health Research; Steven Goldstein, PhD, Study Chair — University of Michigan Henry Ruppenthal Family Professor of Orthopaedic Surgery and Bioengineering
Locations (1):
- University of Michigan Center for Oral Health Research, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Albrektsson T, Branemark PI, Hansson HA, Lindstrom J. Osseointegrated titanium implants. Requirements for ensuring a long-lasting, direct bone-to-implant anchorage in man. Acta Orthop Scand. 1981;52(2):155-70. doi: 10.3109/17453678108991776. PMID 7246093
- [Background] Albrektsson T, Lekholm U. Osseointegration: current state of the art. Dent Clin North Am. 1989 Oct;33(4):537-54. PMID 2680652
- [Background] Amler MH. The time sequence of tissue regeneration in human extraction wounds. Oral Surg Oral Med Oral Pathol. 1969 Mar;27(3):309-18. doi: 10.1016/0030-4220(69)90357-0. No abstract available. PMID 5251474
- [Background] Atwood DA. Reduction of residual ridges: a major oral disease entity. J Prosthet Dent. 1971 Sep;26(3):266-79. doi: 10.1016/0022-3913(71)90069-2. No abstract available. PMID 4934947
- [Background] Atwood DA, Coy WA. Clinical, cephalometric, and densitometric study of reduction of residual ridges. J Prosthet Dent. 1971 Sep;26(3):280-95. doi: 10.1016/0022-3913(71)90070-9. No abstract available. PMID 5284182
- [Background] Caldwell J, Palsson BO, Locey B, Emerson SG. Culture perfusion schedules influence the metabolic activity and granulocyte-macrophage colony-stimulating factor production rates of human bone marrow stromal cells. J Cell Physiol. 1991 May;147(2):344-53. doi: 10.1002/jcp.1041470221. PMID 2040665
- [Background] Cardaropoli G, Araujo M, Hayacibara R, Sukekava F, Lindhe J. Healing of extraction sockets and surgically produced - augmented and non-augmented - defects in the alveolar ridge. An experimental study in the dog. J Clin Periodontol. 2005 May;32(5):435-40. doi: 10.1111/j.1600-051X.2005.00692.x. PMID 15842256
- [Background] Cardaropoli G, Araujo M, Lindhe J. Dynamics of bone tissue formation in tooth extraction sites. An experimental study in dogs. J Clin Periodontol. 2003 Sep;30(9):809-18. doi: 10.1034/j.1600-051x.2003.00366.x. PMID 12956657
- [Background] Carlsson L, Rostlund T, Albrektsson B, Albrektsson T, Branemark PI. Osseointegration of titanium implants. Acta Orthop Scand. 1986 Aug;57(4):285-9. doi: 10.3109/17453678608994393. PMID 3788488
- [Background] Cochran D. Implant therapy I. Ann Periodontol. 1996 Nov;1(1):707-91. doi: 10.1902/annals.1996.1.1.707. No abstract available. PMID 9118278
- [Background] Colter DC, Class R, DiGirolamo CM, Prockop DJ. Rapid expansion of recycling stem cells in cultures of plastic-adherent cells from human bone marrow. Proc Natl Acad Sci U S A. 2000 Mar 28;97(7):3213-8. doi: 10.1073/pnas.97.7.3213. PMID 10725391
- [Background] De Kok IJ, Drapeau SJ, Young R, Cooper LF. Evaluation of mesenchymal stem cells following implantation in alveolar sockets: a canine safety study. Int J Oral Maxillofac Implants. 2005 Jul-Aug;20(4):511-8. PMID 16161734
- [Background] Evian CI, Rosenberg ES, Coslet JG, Corn H. The osteogenic activity of bone removed from healing extraction sockets in humans. J Periodontol. 1982 Feb;53(2):81-5. doi: 10.1902/jop.1982.53.2.81. PMID 6950085
- [Background] Fiorellini JP, Howell TH, Cochran D, Malmquist J, Lilly LC, Spagnoli D, Toljanic J, Jones A, Nevins M. Randomized study evaluating recombinant human bone morphogenetic protein-2 for extraction socket augmentation. J Periodontol. 2005 Apr;76(4):605-13. doi: 10.1902/jop.2005.76.4.605. PMID 15857102
- [Background] Friedenstein AJ, Ivanov-Smolenski AA, Chajlakjan RK, Gorskaya UF, Kuralesova AI, Latzinik NW, Gerasimow UW. Origin of bone marrow stromal mechanocytes in radiochimeras and heterotopic transplants. Exp Hematol. 1978 May;6(5):440-4. PMID 350596
- [Background] Fugazzotto PA. Success and failure rates of osseointegrated implants in function in regenerated bone for 72 to 133 months. Int J Oral Maxillofac Implants. 2005 Jan-Feb;20(1):77-83. PMID 15747677
- [Background] Gao J, Dennis JE, Solchaga LA, Awadallah AS, Goldberg VM, Caplan AI. Tissue-engineered fabrication of an osteochondral composite graft using rat bone marrow-derived mesenchymal stem cells. Tissue Eng. 2001 Aug;7(4):363-71. doi: 10.1089/10763270152436427. PMID 11506726
- [Background] Iasella JM, Greenwell H, Miller RL, Hill M, Drisko C, Bohra AA, Scheetz JP. Ridge preservation with freeze-dried bone allograft and a collagen membrane compared to extraction alone for implant site development: a clinical and histologic study in humans. J Periodontol. 2003 Jul;74(7):990-9. doi: 10.1902/jop.2003.74.7.990. PMID 12931761
- [Background] Ishaug-Riley SL, Crane GM, Gurlek A, Miller MJ, Yasko AW, Yaszemski MJ, Mikos AG. Ectopic bone formation by marrow stromal osteoblast transplantation using poly(DL-lactic-co-glycolic acid) foams implanted into the rat mesentery. J Biomed Mater Res. 1997 Jul;36(1):1-8. doi: 10.1002/(sici)1097-4636(199707)36:13.0.co;2-p. PMID 9212383
- [Background] Jeffcoat MK, Reddy MS. Advances in measurements of periodontal bone and attachment loss. Monogr Oral Sci. 2000;17:56-72. doi: 10.1159/000061636. PMID 10949835
- [Background] Kaigler D, Krebsbach PH, Wang Z, West ER, Horger K, Mooney DJ. Transplanted endothelial cells enhance orthotopic bone regeneration. J Dent Res. 2006 Jul;85(7):633-7. doi: 10.1177/154405910608500710. PMID 16798864
- [Background] Kaigler D, Mooney D. Tissue engineering's impact on dentistry. J Dent Educ. 2001 May;65(5):456-62. PMID 11425250
- [Background] Krebsbach PH, Kuznetsov SA, Bianco P, Robey PG. Bone marrow stromal cells: characterization and clinical application. Crit Rev Oral Biol Med. 1999;10(2):165-81. doi: 10.1177/10454411990100020401. PMID 10759420
- [Background] Krebsbach PH, Kuznetsov SA, Satomura K, Emmons RV, Rowe DW, Robey PG. Bone formation in vivo: comparison of osteogenesis by transplanted mouse and human marrow stromal fibroblasts. Transplantation. 1997 Apr 27;63(8):1059-69. doi: 10.1097/00007890-199704270-00003. PMID 9133465
- [Background] Langer R, Vacanti JP. Tissue engineering. Science. 1993 May 14;260(5110):920-6. doi: 10.1126/science.8493529.
- [Background] Lekovic V, Camargo PM, Klokkevold PR, Weinlaender M, Kenney EB, Dimitrijevic B, Nedic M. Preservation of alveolar bone in extraction sockets using bioabsorbable membranes. J Periodontol. 1998 Sep;69(9):1044-9. doi: 10.1902/jop.1998.69.9.1044. PMID 9776033
- [Background] Mankani MH, Kuznetsov SA, Wolfe RM, Marshall GW, Robey PG. In vivo bone formation by human bone marrow stromal cells: reconstruction of the mouse calvarium and mandible. Stem Cells. 2006 Sep;24(9):2140-9. doi: 10.1634/stemcells.2005-0567. Epub 2006 Jun 8. PMID 16763200
- [Background] Marei MK, Nouh SR, Saad MM, Ismail NS. Preservation and regeneration of alveolar bone by tissue-engineered implants. Tissue Eng. 2005 May-Jun;11(5-6):751-67. doi: 10.1089/ten.2005.11.751. PMID 15998216
- [Background] Misch CE. Bone classification, training keys to implant success. Dent Today. 1989 May;8(4):39-44. No abstract available. PMID 2597401
- [Background] Nevins M, Giannobile WV, McGuire MK, Kao RT, Mellonig JT, Hinrichs JE, McAllister BS, Murphy KS, McClain PK, Nevins ML, Paquette DW, Han TJ, Reddy MS, Lavin PT, Genco RJ, Lynch SE. Platelet-derived growth factor stimulates bone fill and rate of attachment level gain: results of a large multicenter randomized controlled trial. J Periodontol. 2005 Dec;76(12):2205-15. doi: 10.1902/jop.2005.76.12.2205. PMID 16332231
- [Background] Pecora AL, Stiff P, Jennis A, Goldberg S, Rosenbluth R, Price P, Goltry KL, Douville J, Armstrong RD, Smith AK, Preti RA. Prompt and durable engraftment in two older adult patients with high risk chronic myelogenous leukemia (CML) using ex vivo expanded and unmanipulated unrelated umbilical cord blood. Bone Marrow Transplant. 2000 Apr;25(7):797-9. doi: 10.1038/sj.bmt.1702222. PMID 10745268
- [Background] Pecora AL, Stiff P, LeMaistre CF, Bayer R, Bachier C, Goldberg SL, Parthasarathy M, Jennis AA, Smith AK, Douville J, Chen B, Armstrong RD, Mandalam RK, Preti R. A phase II trial evaluating the safety and effectiveness of the AastromReplicell system for augmentation of low-dose blood stem cell transplantation. Bone Marrow Transplant. 2001 Aug;28(3):295-303. doi: 10.1038/sj.bmt.1703137. PMID 11535999
- [Background] Prockop DJ, Azizi SA, Colter D, Digirolamo C, Kopen G, Phinney DG. Potential use of stem cells from bone marrow to repair the extracellular matrix and the central nervous system. Biochem Soc Trans. 2000;28(4):341-5. PMID 10961915
- [Background] Reynolds MA, Aichelmann-Reidy ME, Branch-Mays GL, Gunsolley JC. The efficacy of bone replacement grafts in the treatment of periodontal osseous defects. A systematic review. Ann Periodontol. 2003 Dec;8(1):227-65. doi: 10.1902/annals.2003.8.1.227. PMID 14971256
- [Background] Schenk RK, Buser D, Hardwick WR, Dahlin C. Healing pattern of bone regeneration in membrane-protected defects: a histologic study in the canine mandible. Int J Oral Maxillofac Implants. 1994 Jan-Feb;9(1):13-29. PMID 8150509
- [Background] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475
- [Background] Schwartz RM, Palsson BO, Emerson SG. Rapid medium perfusion rate significantly increases the productivity and longevity of human bone marrow cultures. Proc Natl Acad Sci U S A. 1991 Aug 1;88(15):6760-4. doi: 10.1073/pnas.88.15.6760. PMID 1862099
- [Background] Seo BM, Miura M, Gronthos S, Bartold PM, Batouli S, Brahim J, Young M, Robey PG, Wang CY, Shi S. Investigation of multipotent postnatal stem cells from human periodontal ligament. Lancet. 2004 Jul 10-16;364(9429):149-55. doi: 10.1016/S0140-6736(04)16627-0. PMID 15246727
- [Background] Shang Q, Wang Z, Liu W, Shi Y, Cui L, Cao Y. Tissue-engineered bone repair of sheep cranial defects with autologous bone marrow stromal cells. J Craniofac Surg. 2001 Nov;12(6):586-93; discussion 594-5. doi: 10.1097/00001665-200111000-00017. PMID 11711828
- [Background] Stanford CM. Bone quantity and quality: are they relevant predictors of implant outcomes? Int J Prosthodont. 2003;16 Suppl:43-5; discussion 47-51. No abstract available. PMID 14661708
- [Background] Taba M Jr, Jin Q, Sugai JV, Giannobile WV. Current concepts in periodontal bioengineering. Orthod Craniofac Res. 2005 Nov;8(4):292-302. doi: 10.1111/j.1601-6343.2005.00352.x. PMID 16238610
- [Background] Wang Z, Song J, Taichman RS, Krebsbach PH. Ablation of proliferating marrow with 5-fluorouracil allows partial purification of mesenchymal stem cells. Stem Cells. 2006 Jun;24(6):1573-82. doi: 10.1634/stemcells.2005-0399. PMID 16769762
- [Background] Wenzel A. Bitewing and digital bitewing radiography for detection of caries lesions. J Dent Res. 2004;83 Spec No C:C72-5. doi: 10.1177/154405910408301s14. PMID 15286126
- [Derived] Kaigler D, Pagni G, Park CH, Braun TM, Holman LA, Yi E, Tarle SA, Bartel RL, Giannobile WV. Stem cell therapy for craniofacial bone regeneration: a randomized, controlled feasibility trial. Cell Transplant. 2013;22(5):767-77. doi: 10.3727/096368912X652968. PMID 22776413

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Subjects will receive Tissue Repair Cell (TRC) therapy plus Gelfoam carrier
Period: Overall Study
Arm/Group | Treatment | Control
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (11) | 53 (14) | 50 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Bone Regeneration
Description: The primary objective of this study is to determine whether the placement of Tissue Repair Cells (TRCs) at the time of tooth extraction can safely and effectively promote bone regeneration in alveolar bone defects created by tooth extraction.
  * Safety was assessed through adverse event reporting
  * Bone regeneration was assessed through measures of bone mineral density and bone volume fraction of biopsied regenerated bone tissue. Bone regeneration was also measured through radiographic analysis of relative bone height gain (% of the bone height regenerated relative to the height before tooth extraction)
Time Frame: 12 months after tooth extraction
Measure: Mean (Standard Deviation); unit: % bone height
Arm/Group | Tissue Repair Cells (TRC) | Control
Number analyzed (Participants) | 12 | 12
% bone height | 79 (10) [6 to 4] | 63 (16)

2. Secondary Outcome: Number of Participants Who Successfully Received Dental Implant Fixtures
Description: The secondary objective is to determine if Tissue Repair Cell therapy regenerates bone enabling the installation and stability of dental implant fixtures
Time Frame: 12 months after tooth extraction
Measure: Number; unit: participants
Arm/Group | Tissue Repair Cells (TRC) | Control
Number analyzed (Participants) | 12 | 12
participants | 12 | 12

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Experimental: Tissue Repair Cell (TRC): Subjects will receive TRC therapy plus Gelfoam carrier
- Sham Comparator: Control: Subjects will receive the control treatment, consisting of Gelfoam carrier without Tissue Repair Cell (TRC) therapy.
Arm/Group | Experimental: Tissue Repair Cell (TRC) | Sham Comparator: Control
Serious Adverse Events (participants affected / at risk) | 0/12 | 3/12
Other Adverse Events (participants affected / at risk) | 10/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Tissue Repair Cell (TRC) (N=12) | Sham Comparator: Control (N=12)
Stomach Ulcer (Surgical and medical procedures) | 0 (0) | 1 (1) — Hospitalized for 19 days.
Assault injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Hospitalized for 2-3 days.
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Hospitalized 3 days
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Experimental: Tissue Repair Cell (TRC) (N=12) | Sham Comparator: Control (N=12)
Soreness following aspiration (Surgical and medical procedures) | 1 (1) | 0 (0)
Anxiety prior to procedure (Social circumstances) | 1 (1) | 0 (0)
Post extraction soreness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pulled leg muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fractured tooth (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Discomfort near surgical site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Restoration defect (Surgical and medical procedures) | 1 (1) | 0 (0)
Upper lip tingling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Oral conidition requiring multiple extractions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fractured tooth (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Post surgical infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Shingles (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flu (General disorders) | 0 (0) | 1 (1)
Dislocated knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Swelling and tenderness in tooth extraction area (Surgical and medical procedures) | 0 (0) | 1 (1)
Fractured tooth extracted (Surgical and medical procedures) | 0 (0) | 1 (1)
Sensitive tooth (Nervous system disorders) | 0 (0) | 1 (1)
Post extraction pain (Surgical and medical procedures) | 0 (0) | 1 (1)
Open incision due to sutures coming out (Surgical and medical procedures) | 1 (1) | 0 (0)
Discomfort with mouth movement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Slight incision opening (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Slight incision opening (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pressure in sinus following extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Fractured teeth extracted (Surgical and medical procedures) | 1 (1) | 0 (0)
Non-restorable tooth extracted (Surgical and medical procedures) | 1 (1) | 0 (0)
Distress from theft (Nervous system disorders) | 0 (0) | 1 (1)
Swelling and oozing following extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Slight incision opening (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Discomfort (Surgical and medical procedures) | 0 (0) | 1 (1)
Fractured tooth extracted (Surgical and medical procedures) | 0 (0) | 1/1 (1)
Slight incision opening (Skin and subcutaneous tissue disorders) | 0 (0) | 1/1 (1)
Non-restorable tooth extracted (Surgical and medical procedures) | 0 (0) | 1 (1)
Implant cover screw fell out and was replaced (Surgical and medical procedures) | 0 (0) | 1 (1)
Fractured tooth extracted (Surgical and medical procedures) | 1 (1) | 0 (0)
Failed aspiration (Surgical and medical procedures) | 1 (1) | 0 (0)
Bruising aspiration site (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Moderate-severe swelling following extraction (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mild swelling and bruising following extraction (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fractured tooth (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Non-restorable teeth extracted (Surgical and medical procedures) | 0 (0) | 1 (1)
Moderate bruising and swelling following implant uncovery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Supporation from tip of nose (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Crown fell off (Surgical and medical procedures) | 0 (0) | 1 (1)
Broken upper flipper (Surgical and medical procedures) | 0 (0) | 1 (1)
Cut tendon in hand (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fell down stairs and tore tendons in right foot (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-op bleeding at aspiration site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Relocated to another state due to personal issues (Social circumstances) | 1 (1) | 0 (0)
Implant cover screw fell out (Surgical and medical procedures) | 1 (1) | 0 (0)
Pink eye (Eye disorders) | 1 (1) | 0 (0)
Bruising following extraction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fractured tooth (Surgical and medical procedures) | 1 (1) | 0 (0)
Tissue near extaction site loose causing some tenderness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Soreness in extraction site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Choking while eating (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute pharyngitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — PCP
Strep throat (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Swelling following extraction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bruising following extraction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Discomfort following implant uncovery (Surgical and medical procedures) | 0 (0) | 1 (1)
Post-op bleeding at aspiration site (Surgical and medical procedures) | 1 (1) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Post-op bleeding at aspiration site (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bruising and swelling following extraction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bone exposure following extraction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — non-study area
Sensitivity to sweet and cold (Nervous system disorders) | 1 (1) | 0 (0)
Swelling following extraction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nausea from medication (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain and leg cramping during aspiration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured teeth extracted (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical treatment for addiction (Surgical and medical procedures) | 1 (1) | 0 (0)
Crown fell off (Surgical and medical procedures) | 0 (0) | 1 (1)
Broken flipper (Surgical and medical procedures) | 1 (1) | 0 (0)
Acute pharyngitis (General disorders) | 0 (0) | 1 (1) — ER
Density in lungs (General disorders) | 0 (0) | 1 (1)
Failed aspiration (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes